CLINICAL TRIAL: NCT06689787
Title: A Mobile Health Intervention to Improve Psychosocial Functioning in Veterans With Posttraumatic Stress Disorder and Depression Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D5318-W; IK2RX005318-01A1 (NIH)
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Psychosocial Functioning; Stress Disorders, Post-Traumatic; Depressive Disorder, Major
Keywords: Veterans; Mobile Applications
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-Guided STAIR Coach with Real-Time Assessment (Experimental): Participants randomized to this condition will receive two mobile apps.
  Interventions: Other: Self-Guided STAIR Coach with Real-Time Assessment
- Real-Time Assessment (Active Comparator): Participants randomized to this condition will receive one mobile app.
  Interventions: Other: Real-Time Assessment

INTERVENTIONS:
Other: Self-Guided STAIR Coach with Real-Time Assessment — Two mobile apps to be used as one intervention package to support participants in their progress through STAIR (Skills Training in Affective and Interpersonal Regulation) with self-monitoring of symptoms and functioning
  Arms: Self-Guided STAIR Coach with Real-Time Assessment
Other: Real-Time Assessment — One mobile app to support participants in self-monitoring of symptoms and functioning
  Arms: Real-Time Assessment

SUMMARY:
Posttraumatic stress disorder (PTSD) and depression are the two most common mental health conditions among Veterans. When Veterans experience both, there is a negative impact on their functioning, making it difficult to function at work or at home and socially with other people. Although talk therapies can result in improvements in functioning, they are difficult to access because there are limited clinicians who can provide them. As most US adults now own a smartphone, mobile apps are a way for Veterans to access content traditionally delivered through talk therapies at their own pace. This study will test a mobile app based on a trauma-informed talk therapy that has helped Veterans with PTSD and depression make large improvements in functioning, through learning skills to navigate emotions and relationships. Additionally, through answering brief surveys and enabling passive tracking on their smartphones, Veterans will see real-time information on their functioning and mental health and on potential benefits from using these skills.

DETAILED DESCRIPTION:
Veterans experience high rates of posttraumatic stress disorder (PTSD) and depression, which are frequently comorbid and result in difficulties with psychosocial functioning substantially greater than either disorder alone. Functioning difficulties in Veterans have not been adequately addressed by most existing psychotherapies for PTSD and depression because they often focus on symptom improvement and are highly resource-intensive, requiring the training and time of skilled providers. To address this gap, mobile health (mHealth) apps can serve as a widely accessible, standalone or adjunctive intervention to target psychosocial functioning among Veterans with comorbid PTSD and depression. This study focuses on the evaluation of a self-guided mHealth intervention based on Skills Training in Affective and Interpersonal Regulation (STAIR), an evidence-based psychotherapy that explicitly targets functioning improvements and also alleviates PTSD and depression symptoms among trauma survivors. As part of the intervention, real-time assessment (i.e., ecological momentary assessment and passive sensing) will be incorporated to support Veterans in monitoring their functioning, symptoms, and potential benefits from STAIR. The primary goal is to determine the feasibility and acceptability of this intervention (self-guided STAIR Coach with real-time assessment).

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* enrolled in VA care
* fluent in English
* able to provide informed consent
* own a smartphone or willing to use a study-provided smartphone
* have diagnoses of current posttraumatic stress disorder (PTSD) and major depressive disorder (MDD)
* willing to not begin another form of Skills Training in Affective and Interpersonal Regulation (STAIR) during the study

Exclusion Criteria:

* history of mania or psychosis
* current suicidal ideation with plan and intent to harm self
* acute intoxication from alcohol or other substances
* current or past experience with any form of STAIR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2027-04-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Study Recruitment Rate | Evaluated at end of trial (lasting approximately 2 years)
  Recruitment rate will be calculated as the number of participants who are eligible for the study divided by the number of screened participants. Target feasibility benchmark is 50%.
Study Retention Rate | Evaluated at end of trial (lasting approximately 2 years)
  Retention rate will be calculated as the number of participants who completed the full study divided by the total number of enrolled participants. Target feasibility benchmark is 70%.
Study Engagement Rate | Evaluated at end of trial (lasting approximately 2 years)
  Engagement rate will refer to the mean percentage of completed STAIR Coach training plan levels and completed EMA surveys. Target feasibility benchmark is 70%.
Mobile Application Rating Scale User Version (uMARS) | Post-treatment (i.e., 12 weeks after starting the trial)
  App quality will be assessed through the Mobile Application Rating Scale User Version (uMARS). Total scores on the uMARS range from 1 to 5, with higher scores indicating higher quality. Target acceptability benchmark is a uMARS mean score of greater than or equal to 4 (indicating positive app quality).
Client Satisfaction Questionnaire-8 (CSQ-8) | Post-treatment (i.e., 12 weeks after starting the trial)
  Client satisfaction will be assessed through the Client Satisfaction Questionnaire-8 (CSQ-8). Total scores on the CSQ-8 range from 8 to 32, with higher scores indicating higher satisfaction. Acceptability benchmark is a CSQ-8 mean score of greater than or equal to 24 (indicating general treatment satisfaction).

SECONDARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Baseline, midpoint, post-treatment, follow-up (i.e., 0 weeks, 6 weeks, 12 weeks, and 18 weeks after starting the trial, respectively)
  PTSD symptoms will be assessed through the PTSD Checklist for DSM-5 (PCL-5). Total scores on the PCL-5 range from 0 to 80, with higher scores indicating greater PTSD symptoms. The focus will be on evaluating effect sizes and not statistical significance. Effect sizes will be inspected to see whether they are in the expected direction and larger for the intervention condition compared to the control condition.
Patient Health Questionnaire-9 (PHQ-9) | Baseline, midpoint, post-treatment, follow-up (i.e., 0 weeks, 6 weeks, 12 weeks, and 18 weeks after starting the trial, respectively)
  Depression symptoms will be assessed through the Patient Health Questionnaire-9 (PHQ-9). Total scores on the PHQ-9 range from 0 to 27, with higher scores indicating greater depression symptoms. The focus will be on evaluating effect sizes and not statistical significance. Effect sizes will be inspected to see whether they are in the expected direction and larger for the intervention condition compared to the control condition.
World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | Baseline, midpoint, post-treatment, follow-up (i.e., 0 weeks, 6 weeks, 12 weeks, and 18 weeks after starting the trial, respectively)
  Psychosocial functioning impairment will be assessed through the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0). Total scores on the WHODAS 2.0 range from 0 to 144, with higher scores indicating greater functioning impairment. The focus will be on evaluating effect sizes and not statistical significance. Effect sizes will be inspected to see whether they are in the expected direction and larger for the intervention condition compared to the control condition.

CONTACTS AND LOCATIONS:
Overall Officials: Haijing Wu Hallenbeck, PhD MA, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No